CLINICAL TRIAL: NCT02947581
Title: A Randomized Trial of Combined Albendazole Plus Praziquantel for Subarachnoid Cysticercosis of the Sylvian Fissure or the Basal Cisterns
Brief Title: Sub Arachnoid Neurocysticercosis Treatment Outcome (SANTO)
Acronym: SANTO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Albendazole and albendazole placebo are not available in our local suppliers or in the international market. Consequently, it is no possible to re-initiate the enrollment to complete the original sample size.
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61449
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Neurocysticercosis
Keywords: subarachnoid neurocysticercosis; albendazole; praziquantel
MeSH Terms: conditions — Neurocysticercosis | interventions — Albendazole; Praziquantel

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled study in patients with subarachnoid cysticercosis of the basal cisterns or the Sylvian fissure, comparing in two parallel arms the efficacy of the standard of care anti-parasitic regime (30 days of ABZ at 15 mg/k/d, up to 1200 mg/k/d) with a combined regime using similar doses of ABZ and adding PZQ at 50 mg/k/d for the initial 15 days of anti-parasitic treatment. The study and interim analysis plan are designed to allow direct, concrete efficacy comparison in this deadly type of NCC while minimizing the risks of disease progression in the standard of care arm.
Who Masked: Participant, Investigator
Masking Description: Tablets containing placebo for PZQ and placebo for ABZ will be purchased from the same commercial sources than those containing active drug if possible. As much as possible, they should have the same size, appearance, excipient, smell, and taste as those containing active drug. A preliminary evaluation of the potential for distinction of active drug and placebo by patients will be performed by the investigators before randomization of the drugs and placebos to their individual coded packages. If distinguishable, a new lot will be ordered.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventions (Experimental): Albendazole and praziquantel. Albendazole: 15 mg/k/d up to 800 mg/d (days 1 to 20), followed by 15 mg/k/d up to 1200 mg/d (day 21 to 30) and prazicuantel (50 mg/k/d days 1 to 15).
  Interventions: Drug: Albendazole and praziquantel
- Comparison regime (Active Comparator): Albendazole and praziquantel placebo. Albendazole: 15 mg/k/d (days 1 to 30) and prazicuantel placebo in similar doses 50 mg/k/d (days 1 to 15).
  Interventions: Drug: Albendazole and praziquantel placebo

INTERVENTIONS:
Drug: Albendazole and praziquantel — Intervention - PZQ (50 mg/k/d, up to 3600 mg/d, for 15 days), as an add-on to ABZ treatment (15 mg/k/d, up to 800 mg/d for days 1-20, up to 1200 mg/d for days 21-30). In order to maintain the double blind nature of the trial, ABZ placebo will be administered to individuals over 53 kg of weight until completing the equivalent doses in the comparison group.
  Other Names: ABZ+PZQ
  Arms: Interventions
Drug: Albendazole and praziquantel placebo — PZQ placebo in similar doses, given during the initial 15 days of ABZ treatment at standard doses (15 mg/k/d up to 1200 mg/d for 30 days)
  Other Names: ABZ+PZQ PCB
  Arms: Comparison regime

SUMMARY:
Taenia solium neurocysticercosis (NCC) is a parasitic infection causing much neurological disease in most of the world. When parasites locate in the cavities around the brain (subarachnoid NCC, SANCC), it becomes an aggressive, progressive and frequently lethal presentation. Current treatment regimens for SANCC have quite limited efficacy. The investigators propose to compare the current standard of care (a single antiparasitic drug, albendazole) with a combined regimen using two antiparasitic drugs simultaneously by adding praziquantel. The trial will enrol 164 patients in four centers, two in Peru, one in Ecuador, and one in Brasil.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled study in patients with subarachnoid cysticercosis of the basal cisterns or the Sylvian fissure, comparing in two parallel arms the efficacy of the standard of care anti-parasitic regime (30 days of ABZ at 15 mg/k/d, up to 1200 mg/k/d) with a combined regime using similar doses of ABZ and adding PZQ at 50 mg/k/d for the initial 15 days of anti-parasitic treatment. The study and interim analysis plan are designed to allow direct, concrete efficacy comparison in this deadly type of NCC while minimizing the risks of disease progression in the standard of care arm.

In short, this is a parallel group study with a dichotomous primary outcome variable. The main analysis will compare the proportions of patients obtaining the primary outcome at 6 months, using a Chi-square test in a bivariate analysis. A similar analysis will be used for the proportions of patients with a good clinical outcome, and the proportions of patients in whom lesion resolution sustains when assessed at month 12. A Student T test analysis will be used to compare for reduction in parasite volume and non-parametric Mann-Whitney test will be alternatively applied for non-normally distributed data. A non-parametric Spearman's Rho test will be used to assess the correlation between the proportions of cyst mass reduction with the decrease in antigen levels in each study group. A Chi-square test in a bivariate analysis will evaluate the association between negative antigen levels at 6 months versus the complete disappearance of cyst mass.

ELIGIBILITY:
Inclusion Criteria:

* - Male or female adult individuals (18 to 65 y.o.) with a diagnosis of basal subarachnoid cysticercosis (including locations in the Sylvian fissure or lower interhemispheric spaces) by neuroimaging and confirmed by serology.
* Baseline laboratory results along acceptable ranges (specifically defined in the study protocol).
* Willingness to accomplish the two-week minimum hospitalization required.

Exclusion Criteria:

* Previous therapy with ABZ or PZQ in the preceding 3 years (except for patients who received single-dose ABZ for intestinal parasites, or patients who received antiparasitic treatment between one and three years before enrollment but demonstrated lesion persistence or progression during the past 12 months).
* A type of NCC which can expose the patient to increased risk during the study, specifically: a) intraventricular cysts; b) cysts in brainstem; c) concomitant intraparenchymal lesions greater than 3 cm of diameter in addition to their SANCC lesions; d) more than 20 intraparenchymal cysts in addition to their SANCC lesions; or d) untreated ocular cysticercosis. Patients with a lateral ventricle cyst, less than 2 cm in diameter, without hydrocephalus or intracranial hypertension, can be included. The presence of concomitant intraparenchymal cysts of less than 3 cm in diameter will not exclude the patient unless there are more than 20 of them.
* Active pulmonary tuberculosis evidenced by positive chest X-ray and positive sputum smears, or symptoms compatible with tuberculosis (fever+sweats or fever+cough) not otherwise explained.
* Individuals with positive markers for active hepatitis.
* Systemic disease that may affect therapy or short-term prognosis, including but not limited to chronic renal failure, hepatic insufficiency, cardiac failure, and steroid-dependent immune diseases.
* Patients in unstable condition or with symptomatic intracranial hypertension (ICH). Definition of symptomatic ICH for this study is the presence of headaches, nausea, and vomiting, with papilledema at fundoscopic examination. Patients in this category can be considered for entrance into the study only after resolution of ICH by ventricular-peritoneal shunting or neuroendoscopic procedures involving CSF flow derivation. These procedures would be done as part of their standard medical care and are not part of the trial intervention.
* Pregnancy during anti-parasitic treatment. If a patient becomes pregnant after treatment, she will continue in the study but will have radiological exams delayed until after delivery.
* History of hypersensitivity to ABZ or PZQ
* Chronic or drug abuse as defined in the study protocol.
* Unwilling or unable to undergo MRI exams (like patients with ferromagnetic implants)
* Inability or unwillingness of subject or legal representative to give written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
Radiological efficacy at three months (3-month improvement). | Day 90 +/- 15 days
  Thirty percent or greater decrease in the combined volume of all parasitic masses, evaluated by contrast-enhanced MRI 3 months after therapy onset, and recorded both as a dichotomous outcome and as a continuous quantification.

SECONDARY OUTCOMES:
Radiological efficacy at six months (marked improvement or "radiological cure") (evaluated only in patients with improvement at month 3). | Day 180 +/- 15 days
  Total disappearance or greater than 50% decrease in the combined volume of subarachnoid parasites, evaluated by contrast-enhanced MRI 6 months after therapy onset, and recorded both as a dichotomous outcome and as a continuous quantification. three.months after treatment onset (comparative between treatment arms).
Effect persistence at 12 months (no relapse) (evaluated only in patients with marked improvement at month 6) Effect persistence at 12 months (no relapse) (evaluated only in patients with marked improvement at month 6) | Day 365 +/- 15 days
  No reappearance or re-growth of the parasitic lesions on contrast enhanced MRI at 12 months after therapy onset, recorded as a dichotomous outcome. hypertension, or progressive neurologic deficits (in cognitive functions, motor function, gait, or other defined neurological signs) in a patient off steroid therapy, as assessed by a study neurologist 12 months post treatment.
Clinically asymptomatic patient | 3, 6, and 12 months
  No evidence of uncontrolled seizures, chronic severe headaches, intracranial hypertension, or progressive neurologic deficits (in cognitive functions, motor function, gait, or other defined neurological signs) in a patient off steroid therapy, as assessed by a study neurologist at 3, 6, and 12 months post treatment.
Decrease in serum levels | 3 months
  will be measured at 3 months, and expressed as a proportion of the baseline level. This variable will be compared between arms

CONTACTS AND LOCATIONS:
Overall Officials: Hector H. Garcia Lescano, Ph.D, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (2):
- Peru (2):
  - Cysticercosis Unit, Instituto Nacional de Ciencias Neurologicas, Lima
  - Hospital Nacional Cayetano Heredia, Lima

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient data will be shared upon request and review by the project leaders.
Supporting Information: Study Protocol, ICF
Time Frame: Available: December 2021, until December 2023
Access Criteria: The information will be shared upon requested by interested researchers